CLINICAL TRIAL: NCT00131534
Title: The Trauma Recovery and Resiliency Research Project
Status: Completed | Type: Observational
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: CHA-IRB-0031/01/04
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Posttraumatic Stress Disorders
Keywords: Complex trauma; Trauma recovery; Resiliency; Posttraumatic stress; Individual psychotherapy; Group psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychotherapy, Group

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Individual therapy — Stage-based individual therapy for trauma survivors
Behavioral: Group therapy — Stage-based group therapy for trauma survivors

SUMMARY:
The overall purpose of this study is the assessment of treatment outcome among traumatized patients seeking individual and/or group therapy at the Victims of Violence Program. The study gathers information from patients using quantitative (self-report) and qualitative (interview-based) approaches, to determine changes in symptom patterns and domains of functioning relevant to psychological trauma.

DETAILED DESCRIPTION:
The focus of the Trauma Recovery and Resiliency Project is primarily the evaluation of treatment outcome among complexly traumatized patients seeking individual and/or group therapy at the Victims of Violence (VOV) Program, a specialty clinic located in the Outpatient Psychiatry Department of the Cambridge Health Alliance and affiliated with Harvard Medical School. The project has two major components: (1) All patients seeking VOV treatment are administered a battery of self-report measures assessing symptoms associated with complex trauma (i.e., interpersonal trauma that is usually repeated and prolonged) (2) A subsample of patients are interviewed using the Multidimensional Trauma Recovery and Resiliency Interview (MTRRI) and its companion rating scale (MTRR; Harvey et al, 1994, 2000, 2003) to assess trauma impact, recovery and resiliency on eight domains of psychological functioning. Data is analyzed using quantitative and qualitative approaches to evaluate treatment effectiveness and elucidate the recovery trajectories of patients receiving VOV treatment. Two subprojects include (a) preparation of a treatment manual documenting the Women's Trauma Recovery Group, and (b) pilot testing a new interview-based measure of complex trauma symptoms, the Symptoms of Trauma Scale (SOTS).

ELIGIBILITY:
Inclusion Criteria:

* In individual or group therapy at VOV program
* Consents to research participation

Exclusion Criteria:

* Insufficient proficiency in English to complete self-report measures and/or interview
* Research participation clinically counterindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma survivors receiving outpatient treatment.
Sampling Method: Non-Probability Sample
Enrollment: 969 (Actual)
Dates: Start 1991-08; Primary Completion 2009-02 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary R. Harvey, Ph.D., Principal Investigator — Victims of Violence Program, Cambridge Health Alliance; Judith L. Herman, MD, Principal Investigator — Victims of Violence Program, Cambridge Health Alliance; Michaela Mendelsohn, Ph.D., Principal Investigator — Victims of Violence Program, Cambridge Health Alliance
Locations (1):
- Victims of Violence Program, Cambridge Health Alliance, Somerville, Massachusetts, United States

REFERENCES:
- [Background] Harney PA, Harvey MR. Group psychotherapy: An overview. In BH Young & DD Blake (Eds.), Group treatments for post-traumatic stress disorder (pp. 1-13). New York, NY: Brunner/Mazel, 1999.
- [Background] Harvey MR. An ecological view of psychological trauma and trauma recovery. J Trauma Stress. 1996 Jan;9(1):3-23. PMID 8750448
- [Background] Harvey MR, Harney PA. Individual psychotherapy. In C Classen & ID Yalom (Eds.), Treating women molested in childhood (pp. 63-91). San Francisco, CA: Jossey-Bass Publishers, 1995.
- [Background] Harvey MR, Liang B, Harney PA, Koenen K, Tummala-Narra P, Lebowitz L. A multidimensional approach to the assessment of trauma impact, recovery and resiliency: Initial psychometric findings. Journal of Aggression, Maltreatment and Trauma, 6: 87-109, 2003.
- [Background] Harvey MR, Mishler EG, Koenen K, Harney PA. In the aftermath of sexual abuse: Making and remaking meaning in narratives of trauma and recovery. Narrative Inquiry, 10: 291-311, 2000.
- [Background] Harvey MR, Weston D. Multidimensional trauma recovery and resiliency measures: The MTRRI (Interview) and the MTRRQ (Sort). In BH Stamm (Ed.), Measurement of stress, trauma, and adaptation (pp. 209-211). Lutherville, MD: The Sidran Press, 1996.
- [Background] Herman, JL. Complex PTSD: A syndrome in survivors of prolonged and repeated trauma. Journal of Traumatic Stress, 3: 377-391, 1992.
- [Background] Herman JL. Trauma and recovery. New York: Basic Books, 1992.
- [Background] Mendelsohn M, Zachary R, Harney P. Group therapy as an ecological bridge to a new community. Special issue of Journal of Aggression, Maltreatment and Trauma, 14, 227-243.
- [Result] Forman EM, Lynch SM, Bryant TS, Herman JL. Using effectiveness and patient-focused data to evaluate outcome of a community-based trauma treatment. Paper presented at the 17th Annual Meeting of the International Society for Traumatic Stress Studies, New Orleans, LA, 2001.
- [Result] Mendelsohn M, Forman EM, Lynch SM, Herman JL. Group therapy at the Victims of Violence Program: Preliminary Findings. Paper presented at 20th Annual Meeting of the International Society for Traumatic Stress Studies; New Orleans, LA, 2004.
- [Result] Lynch S, Forman E, Mendelsohn M, Herman, JL. A comparison of high and low dissociators' response to trauma-focused treatment. Paper presented at the 21st Conference of the International Society for the Study of Dissociation; New Orleans, LA; 2004.
- [Result] Lynch SM, Forman E, Mendelsohn M, Herman J. Attending to dissociation: assessing change in dissociation and predicting treatment outcome. J Trauma Dissociation. 2008;9(3):301-19. doi: 10.1080/15299730802139063. PMID 19042780
- [Result] Dutra L, Callahan K, Forman E, Mendelsohn M, Herman J. Core schemas and suicidality in a chronically traumatized population. J Nerv Ment Dis. 2008 Jan;196(1):71-4. doi: 10.1097/NMD.0b013e31815fa4c1. PMID 18195645
- [Result] Lynch SM, Keasler AL, Reaves, RC, Channer EG, Bukowski LT. The Story of My Strength: An Exploration of Resilience in the Narratives of Trauma Survivors Early in Recovery. Journal of Aggression, Maltreatment & Trauma 14: 75-97, 2007 Publisher: Haworth Press